CLINICAL TRIAL: NCT00178919
Title: Cardiovascular Regulation: Autonomic/Metabolic Mechanisms PO1 HL56693, Project 4: Cardiovascular Regulation: Autonomic/Metabolic Mechanisms
Brief Title: Nitric Oxide and the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: 010876; NIH 1RO1HL71172
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2010-05-03 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension; Pure Autonomic Failure
Keywords: Endothelial Nitric Oxide; L-NMMA; Trimethaphan; Autonomic Nervous System; Nitric Oxide Inhibition
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure | interventions — omega-N-Methylarginine; Trimethaphan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autonomic Failure Patients (Experimental): To compare the effects of NO inhibition during intact and transient pharmacological blockade of the autonomic nervous system in Patients with Autonomic Failure.
  Interventions: Drug: L-NMMA; Drug: Trimethaphan
- Controls and hypertensives (Experimental): To compare the effects of NO inhibition during intact and transient pharmacological blockade of the autonomic nervous system in normal volunteers and hypertensive subjects.
  Interventions: Drug: L-NMMA; Drug: Trimethaphan

INTERVENTIONS:
Drug: L-NMMA — IV infusion of 125, 250 and 500 mcg/Kg/min for 15 minutes each dose. The main outcome is the maximal increase in blood pressure produced at the end of the infusions or a maximal systolic blood pressure of 160 mm Hg. It could be achieved after the first dose or the third.
Drug: Trimethaphan — IV infusion for the duration of the study at 4-6 mg/min depending on autonomic blockade. This is only to produce transient pharmacological blockade of the autonomic nervous system in order to allow the full expression of the inhibition of nitric oxide synthase. There is no direct outcome associated with this intervention.

SUMMARY:
The amount of blood flowing to the different parts of the body is regulated by the autonomic (automatic) nerves and by local factors produced by the blood vessels. Nitric oxide (NO) is one of the most important of these metabolic factors. If the production of NO is slowed or stopped the amount of blood to the different parts of the body is decreased. There is increasing knowledge that NO mechanisms are impaired in a number of medical conditions. NO function is reduced in patients with risk factors for atherosclerosis (hardening of the arteries) such as hypercholesterolemia (patients with high cholesterol), or diabetes mellitus, and is also impaired in smokers. This NO "deficiency" is believed to contribute to the greater cardiovascular risk that marks these patient populations. This study is designed to examine if endothelial nitric oxide is an important control mechanism of blood pressure under normal conditions, and if impairment of nitric oxide contributes to hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects.
* 18 to 85 years.
* Non-smokers or long term smokers for specific aim 6.
* Drug-free.
* Long term hypertension in specific substudy 3, patients with autonomic failure in specific aims 4 and 5, diabetes mellitus in specific aim 5.

Exclusion Criteria:

* Being on any medication other than antihypertensives (for hypertensives), autonomic medications (for autonomic failure [AF] patients), insulin or other treatment for diabetes (for diabetic patients).
* Having pulmonary, renal, hematopoietic, hepatic and/or cardiac disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Autonomic Dysfunction Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Gamboa A, Shibao C, Diedrich A, Paranjape SY, Farley G, Christman B, Raj SR, Robertson D, Biaggioni I. Excessive nitric oxide function and blood pressure regulation in patients with autonomic failure. Hypertension. 2008 Jun;51(6):1531-6. doi: 10.1161/HYPERTENSIONAHA.107.105171. Epub 2008 Apr 21. PMID 18426998
- [Derived] Gamboa A, Shibao C, Diedrich A, Choi L, Pohar B, Jordan J, Paranjape S, Farley G, Biaggioni I. Contribution of endothelial nitric oxide to blood pressure in humans. Hypertension. 2007 Jan;49(1):170-7. doi: 10.1161/01.HYP.0000252425.06216.26. Epub 2006 Nov 27. PMID 17130304

RESULTS

PARTICIPANT FLOW:
Groups:
- Autonomic Failure Patients: The NO synthase inhibitor L-NMMA was infused intravenously at different doses (125, 250 and 500 mcg/kg/min) until a systolic blood pressure of 150 mm Hg was reached.
- Hypertensives and Controls: The NO synthase inhibitor L-NMMA was infused intravenously at different doses (250, 500 mcg/kg/min) for 15 minutes each dose after acute transient pharmacological blockade of the autonomic nervous system with trimethaphan (4 mg/min) or with the autonomic nervous system intact.
Period: Overall Study
Arm/Group | Autonomic Failure Patients | Hypertensives and Controls
Started | 19 | 93
Completed | 19 | 68
Not Completed | 0 | 25

BASELINE CHARACTERISTICS:
Groups:
- Autonomic Failure Patients; Hypertensives and Controls: To compare the effects of NO inhibition during intact and transient pharmacological blockade of the autonomic nervous system.
- Total: Total of all reporting groups
Arm/Group | Autonomic Failure Patients | Hypertensives and Controls | Total
Number analyzed (Participants) | 19 | 93 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 93 | 106
  >=65 years | 6 | 0 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (10.4) | 37 (11.8) | 41 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 51 | 60
  Male | 10 | 42 | 52
Region of Enrollment [Number; unit: participants]
  United States | 19 | 93 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: L-NMMA (nitric oxide synthase inhibitor) was infused intravenously at different doses for 15 minutes each, after blocking the autonomic nervous system with trimethaphan. The change in systolic blood pressure at the end of the highest tolerated dose is the main outcome. Trimethaphan infused intravenously was used to produce transient blockade of the autonomic nervous system to allow for a full response to nitric oxide inhibition (in the absence of the baroreflex.
Time Frame: At the end of the highest tolerated dose of IV infusion of L-NMMA
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Autonomic Failure Patients | Hypertensives and Controls
Number analyzed (Participants) | 19 | 68
mm Hg | 43 (6.2) | 21 (8.4)

2. Primary Outcome: Systolic Blood Pressure in Response to Systemic Nitric Oxide Inhibition
Description: Systolic blood pressure at the highest tolerated dose of IV infusion of L-NMMA during autonomic nervous system blockade with trimethaphan. Trimethaphan, infused intravenously was used to produce transient blockade of the autonomic nervous system to allow for a full response to nitric oxide inhibition (in the absence of the baroreflex.
Time Frame: End of 15 minutes of infusion of L-NMMA at the highest tolerated dose
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Autonomic Failure Patients | Hypertensives and Controls
Number analyzed (Participants) | 19 | 68
mm Hg | 152 (6.8) | 136 (13.8)

ADVERSE EVENTS:
Arm/Group | Autonomic Failure Patients | Hypertensives and Controls
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/93
Other Adverse Events (participants affected / at risk) | 0/19 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes